CLINICAL TRIAL: NCT02667054
Title: A Phase III Investigation Of Topical Application Of RX0041-002 On Safety And Efficacy In Local (Topical) Anesthesia For Diagnostic Procedures And Surgeries On Or Through The Accessible Mucous Membranes Of The Nasal Cavities
Brief Title: Topical Anesthetic for Procedures Through the Nose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmaceutical Project Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013011
Record Dates: First submitted 2015-04-23; First posted 2016-01-28 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-01

CONDITIONS: Drug Reaction to Analgesic Nos
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active 4% (Active Comparator): One dose of 4mL of RX0041 4% for one day in the mucous membrane prior to a diagnostic or surgical procedure.
  Interventions: Drug: RX0041 4%
- Placebo (Placebo Comparator): One dose of 4mL of RX0041 placebo for one day in the mucous membrane prior to a diagnostic or surgical procedure.
  Interventions: Drug: Placebo
- Active 8% (Active Comparator): One dose of 4mL of RX0041 8% for one day in the mucous membrane prior to a diagnostic or surgical procedure.
  Interventions: Drug: RX0041 8%

INTERVENTIONS:
Drug: RX0041 4% — Anesthetic
  Other Names: Topical Anesthetic
  Arms: Active 4%
Drug: Placebo — Placebo Comparator
  Other Names: Placebo Topical Anesthetic
  Arms: Placebo
Drug: RX0041 8% — Anesthetic
  Other Names: Topical Anesthetic
  Arms: Active 8%

SUMMARY:
To determine if RX0041-002 is a safe and effective topical anesthetic.

DETAILED DESCRIPTION:
This is a phase III single-dose, randomized , placebo and dose-controlled study to evaluate the safety and efficacy of a RX0041-002 topical solution for local anesthesia during diagnostic procedures and surgeries on or through the mucous membranes of the nasal cavities (e.g. nasal/sinus endoscopy, sinusotomy, fracture nasal turbunate(s), lysis intranasal synechia, insertion of nasal septal prosthesis, biopsy intranasal, excision of nasal polyps, excision turbinate(s), removal of foreign body intranasal, septoplasty, sinus debridement).

ELIGIBILITY:
Inclusion Criteria:

1. Is able to understand and comply with protocol requirements, provide written informed consent and HIPPA authorization. Residents of California must also review and sign the California Subject Bill of Rights.
2. Is male or female ≥18 years of age, inclusive, at the time of dosing.
3. Has a predetermined need from a physician for a diagnostic procedure or surgery on or through the nasal mucous membranes of either one or both nostrils.
4. Has the ability to feel pain sensation normally in the anterior nasal septum, as verified by Von Frey 6.10 filament testing.
5. Has the ability to clearly communicate pain and sensation of the anterior nasal septum.
6. Females (if of child-bearing potential and sexually active) and males (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method from the first dose and for 8 days following last dose of study drug. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm, intrauterine device (IUD), condom, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method or withdrawal.

Exclusion Criteria:

1. Has a known allergy to any ester based anesthetics including cocaine HCl, procaine, tetracaine, chloroprocaine, dibucaine, or benzocaine, and/or any other compounds of the drugs and /or devices that are part of this protocol. (Amide based anesthetic allergies are NOT exclusionary. Amide based anesthetics are: Lidocaine, Mepivicaine, Bupivicaine, Levobupivicaine, Ropivicaine, Etidocaine, Prilocaine, and Articaine).
2. Is < Less than 18 years of age.
3. Has previously received study drug during this study.
4. Has a history of abuse of controlled substances, nasal or otherwise, or has damage to the nasal space, that in the opinion of the investigator might interfere with the ability of the subject or investigator to judge analgesia from the study drug.
5. Has participated in an investigational study or received an investigational drug within 30 days preceding the randomization.
6. Is a pregnant or nursing mother.
7. Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy throughout the study, and for women 30 days and men 90 days after the last dose of investigational product in such a manner that the risk of pregnancy and risk to pregnancy is minimized.
8. Suffers from a condition, other than the need for a diagnostic procedure or surgery on or through the nasal mucous membranes, which in the opinion of the Investigator, would compromise the safety of the subject, the quality of the data, or the normal wound healing process.
9. Has severely traumatized mucosa or sepsis in the nasal cavity.
10. Subjects who have experienced a seizure while taking isoniazid (INH), phenothiazines, chlorpromazine, thioridazine, theophylline, or tricyclic antidepressants such as amitriptyline.
11. Use of any analgesic up to 2 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial. This includes NSAIDs such as ibuprofen, diclofenac, indomethacin, sulindac, tolmetin, ketoprofen, flurbiprofen, naprozen, opioids such as codeine, hydrocodone, hydromorphone, morphine, oxycodone and aspirin, or acetaminophen.
12. Use of any SNRIs/SSRIs up to7 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
13. Use of MAO Inhibitor drugs up to14 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
14. Subjects who have experienced a seizure while taking isoniazid (INH), phenothiazines, chlorpromazine, thioridazine, theophylline, or tricyclic antidepressants such as amitriptyline. Has a history of seizure, with the exception of febrile seizures.
15. Has a history of myocardial infarction, coronary artery disease, congestive heart failure, irregular heart rhythm, or uncontrolled hypertensions (defined as an average SBP ≥140 mmHg or an average DBP ≥90 mmHg) or is taking monoamine oxidase inhibitors. Uncontrolled hypertension is defined as systolic blood pressure greater than or equal to 140 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg.
16. Has a known personal or family history of hereditary pseudocholinesterase deficiency. Study participants will be screened by asking about personal or family history of anesthetic reaction, anesthetic death, and previous diagnosis of psuedochloinesterase deficiency in a relative or personally. Subjects identified with pseudocholinesterase deficiency are at risk for delayed recovery with certain anesthetics (e.g. succinylcholine and ester-based anesthetics).
17. Has a known personal or family history of pheochromocytoma. Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (since 10% of these are familial).
18. Has a known personal or family history of adrenal tumor.
19. Has used amphetamines, stimulant prescription and nonprescription products such as catecholamines (direct and indirect acting sympathomimetics), bronchial inhalers containing sympathomimetics (epinephrine or other beta-receptor agonist) or herbal products in the 2 days prior to screening or has a need to use these drugs during the course of the study.
20. Has screening 12-lead ECG findings of any abnormalities. Generally, these are current or prior myocardial ischemia or infarction, dysrhythmia, or risk of serious dysrhythmia (such as prolonged QT interval). An exception to this would be if sinus bradycardia or sinus tachycardia is present, the Investigator must determine whether this finding is clinically relevant and exclusionary
21. Has a positive urine pregnancy test at Screening or Day 1.
22. Has a positive urine test result for drugs of abuse (amphetamines, barbiturates, cannabinoids, cocaine metabolites, opiates and oxycodone) at Screening or Day 1.
23. Hemoglobin < 8.5 g/dl; a one-time retest will be allowed for Hb 8.3-8.4 g/dl.
24. WBC < 3.5 x 103 cells/mcl; a one-time retest will be allowed for WBC 3.3-3.4 x 103 cells/mcl.
25. Platelets < 100 x 103 platelets/mcl; a one-time retest will be allowed for platelets 90-99 x 103 platelets/mcl.
26. Serum Potassium < 3.5 or > 4.5 mEq/L.
27. Serum ALT, AST, and bilirubin not exceeding 2X ULN for the lab's reference values.
28. Is not suitable for entry into the study in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Anesthetized mucous membrane measured using a Von Frey Pain Measure Device | 20 minutes
  Mucous membrane is anesthetized with topical application of RX0041 by insertion of Pain Measure Device (Von Frey)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Goodhead, MSc, Study Director — PPSI
Locations (2):
- United States (2):
  - Aroesty Advocare ENT, Mount Arlington, New Jersey
  - South Carolina ENT, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No
Data will only be submitted to FDA.